CLINICAL TRIAL: NCT03463031
Title: A Double-Blind, Randomized, Parallel-Group Study to Evaluate the Efficacy, Safety and Tolerability of Fixed Dose Combination GSP 301 Nasal Spray Compared With Placebo Nasal Spray in Pediatric Subjects (Aged 6 to Under 12 Years) With Seasonal Allergic Rhinitis (SAR)
Brief Title: Efficacy and Safety of GSP 301 Nasal Spray in Children (Aged 6 to Under 12 Years) With Seasonal Allergic Rhinitis (SAR)
Acronym: GSP 301-305
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Glenmark Specialty S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GSP 301-305
Record Dates: First submitted 2018-03-05; First posted 2018-03-13 (Actual); Results first posted 2019-10-08 (Actual); Last update posted 2019-10-08 (Actual); Status verified 2019-09

CONDITIONS: Seasonal Allergic Rhinitis (SAR)
Keywords: GSP 301 nasal spray for the treatment of Seasonal Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- GSP 301 NS (Experimental): Fixed dose combination of olopatadine hydrochloride 665 μg and mometasone furoate 25 μg NS
  Interventions: Drug: GSP 301 NS
- GSP 301 Placebo NS (Placebo Comparator): GSP 301 Placebo nasal spray
  Interventions: Drug: GSP 301 Placebo NS

INTERVENTIONS:
Drug: GSP 301 NS — 1 spray in each nostril twice daily for 14 days
  Arms: GSP 301 NS
Drug: GSP 301 Placebo NS — 1 spray in each nostril twice daily for 14 days
  Arms: GSP 301 Placebo NS

SUMMARY:
Study to evaluate the efficacy, safety and tolerability of GSP 301 nasal spray (NS) compared with placebo NS in pediatric subjects (aged 6 to under 12 years) with Seasonal Allergic Rhinitis (SAR).

ELIGIBILITY:
Inclusion Criteria:

1. Male and female subjects aged ≥6 to <12 years
2. Clinical history of SAR (at least 2 years) with exacerbations during the study season for the relevant seasonal allergen (e.g., tree/grass pollen)
3. Demonstrated sensitivity to at least 1 seasonal allergen through positive skin prick test within 12 months prior to screening
4. A 12-hour rTNSS value ≥6 out of a possible 12 for the morning assessment at screening
5. Signed informed consent/assent form (subject and parent/caregiver/legal guardian)

Exclusion Criteria:

1. Females of childbearing potential or pregnant
2. Plans to travel outside the known pollen area for the investigational site for 24 hours or longer during the last 7 days of the run-in period.
3. History of anaphylaxis and/or other severe local reaction(s) to skin testing
4. History and evidence of acute or significant chronic sinusitis or chronic purulent post nasal drip
5. Subjects with an active pulmonary disorder or infection.
6. Subjects with posterior subcapsular cataracts or glaucoma

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 446 (Actual)
Dates: Start 2018-03-16 (Actual); Primary Completion 2018-11-14 (Actual); Study Completion 2018-11-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sudeesh Tantry, PhD, Study Director — Glenmark Pharmaceuticals Ltd.
Locations (32):
- United States (32):
  - Glenmark Investigational Site 18, Mission Viejo, California
  - Glenmark Investigational Site 32, Ontario, California
  - Glenmark Investigational Site 30, Paramount, California
  - Glenmark Investigational Site 17, San Diego, California
  - Glenmark Investigational Site 21, Colorado Springs, Colorado
  - Glenmark Investigational Site 13, Marietta, Georgia
  - Glenmark Investigational Site 26, Savannah, Georgia
  - Glenmark Investigational Site 28, Louisville, Kentucky
  - Glenmark Investigational Site 14, Baltimore, Maryland
  - Glenmark Investigational Site 19, Bethesda, Maryland
  - Glenmark Investigational Site 25, Ypsilanti, Michigan
  - Glenmark Investigational Site 12, Columbia, Missouri
  - Glenmark Investigational Site 10, Rolla, Missouri
  - Glenmark Investigational Site 27, Warrensburg, Missouri
  - Glenmark Investigational Site 15, Omaha, Nebraska
  - Glenmark Investigational Site 3, High Point, North Carolina
  - Glenmark Investigational Site 8, Raleigh, North Carolina
  - Glenmark Investigational Site 11, Cincinnati, Ohio
  - Glenmark Investigational Site 29, Cincinnati, Ohio
  - Glenmark Investigational Site 2, Edmond, Oklahoma
  - Glenmark Investigational Site 33, Tulsa, Oklahoma
  - Glenmark Investigational Site 4, Medford, Oregon
  - Glenmark Investigational Site 6, Spartanburg, South Carolina
  - Glenmark Investigational Site 5, Austin, Texas
  - Glenmark Investigational Site 24, Kerrville, Texas
  - Glenmark Investigational Site 1, New Braunfels, Texas
  - Glenmark Investigational Site 7, San Antonio, Texas
  - Glenmark Investigational Site 9, San Antonio, Texas
  - Glenmark Investigational Site 20, Waco, Texas
  - Glenmark Investigational Site 31, Waco, Texas
  - Glenmark Investigational Site 22, Draper, Utah
  - Glenmark Investigational Site 23, Greenfield, Wisconsin

REFERENCES:
- [Derived] Prenner BM, Amar NJ, Hampel FC Jr, Caracta CF, Wu W. Efficacy and safety of GSP301 nasal spray in children aged 6 to 11 years with seasonal allergic rhinitis. Ann Allergy Asthma Immunol. 2022 Nov;129(5):618-626.e2. doi: 10.1016/j.anai.2022.07.029. Epub 2022 Aug 1. PMID 35926824

RESULTS

PARTICIPANT FLOW:
Groups:
- GSP 301 NS: Fixed dose combination of olopatadine hydrochloride 665 μg and mometasone furoate 25 μg NS.
  Intranasal administration, 1 spray in each nostril BID (AM and PM, approximately 12 hours apart) for 14 days
- Placebo NS: GSP 301 Placebo NS. Intranasal administration, 1 spray in each nostril BID (AM and PM, approximately 12 hours apart) for 14 days
Period: Overall Study
Arm/Group | GSP 301 NS | Placebo NS
Started | 225 | 221
Completed | 215 | 216
Not Completed | 10 | 5
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Investigator/Sponsor Decision | 0 | 1
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 4 | 1
Not completed — Use of prohibited medication by subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- GSP 301 NS; Placebo NS: Intranasal administration, 1 spray in each nostril BID (AM and PM, approximately 12 hours apart) for 14 days
- Total: Total of all reporting groups
Arm/Group | GSP 301 NS | Placebo NS | Total
Number analyzed (Participants) | 225 | 221 | 446
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.7 (1.6) | 8.6 (1.7) | 8.7 (1.7)
Age, Customized [Count of Participants; unit: Participants]
  6 - < 9 | 100 | 99 | 199
  9 - < 12 | 125 | 122 | 247
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 99 | 109 | 208
  Male | 126 | 112 | 238
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 67 | 85 | 152
  Not Hispanic or Latino | 158 | 135 | 293
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 5 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 46 | 44 | 90
  White | 168 | 169 | 337
  More than one race | 3 | 2 | 5
  Unknown or Not Reported | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Average AM and PM Subject-reported 12-hour Reflective Total Nasal Symptom Score ( rTNSS) Over the 14-day Treatment Period
Description: The Reflective Total Nasal Symptom Score (rTNSS) was assessed by 12-hour reflective scoring of the severity of four nasal symptoms (rhinorrhea, sneezing, nasal congestion, nasal itching). Scores ranged from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate, causes interference with activities of daily living and/or sleeping). Each of these four nasal symptoms (rhinorrhea, sneezing, nasal congestion, nasal itching) of the rTNSS is rated on a scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe). The four nasal symptoms of the rTNSS is summed. The total score of the rTNSS ranged from 0 to 12.
Time Frame: Baseline and day 14
Population: The Full Analysis Set (FAS) consisted of all subjects who are randomized and received at least 1 dose of IP and had at least 1 post-baseline primary efficacy assessment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GSP 301 NS | Placebo NS
Number analyzed (Participants) | 222 | 219
units on a scale
  Baseline | 8.83 (1.41) | 8.84 (1.66)
  Mean Change from baseline to end of treatment | -2.2 (0.17) | -1.6 (0.18)
Statistical Analysis 1: Comparison: GSP 301 NS vs Placebo NS; Test type: Superiority; p = 0.001, Mixed Models Analysis; Least Square Mean Difference = -0.6, 95% CI 2-sided [-0.9 to -0.2], Standard Error of Mean 0.17

2. Secondary Outcome: Change From Baseline in Average AM and PM Subject-reported 12-hour Instantaneous Total Nasal Symptom Score (iTNSS) Over the 14-day Treatment Period.
Description: The instantaneous Total Nasal Symptom Score (iTNSS) was assessed by instantaneous (ie, an evaluation of the symptom severity just before taking study medication [within 10 minutes]) of four nasal symptoms (rhinorrhea, sneezing, nasal congestion, nasal itching). Scores ranged from 0 (no signs/symptoms evident) to 3 (severe signs/symptoms that is hard to tolerate, causes interference with activities of daily living and/or sleeping). Each of these four nasal symptoms (rhinorrhea, sneezing, nasal congestion, nasal itching) of the iTNSS is rated on a scale from 0 to 3 (0 = none, 1 = mild, 2 = moderate, 3 = severe). The four nasal symptoms of the iTNSS is summed. The total score of the iTNSS ranged from 0 to 12.
Time Frame: Baseline and day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GSP 301 NS | Placebo NS
Number analyzed (Participants) | 222 | 219
units on a scale
  Baseline | 7.89 (1.93) | 7.82 (2.04)
  Mean Change from baseline to end of treatment | -1.8 (0.17) | -1.1 (0.17)
Statistical Analysis 1: Comparison: GSP 301 NS vs Placebo NS; Test type: Superiority; p < 0.001, Mixed Models Analysis; Least Square Mean Difference = -0.6, 95% CI 2-sided [-1.0 to -0.3], Standard Error of Mean 0.17

3. Secondary Outcome: Change From Baseline in the Overall Pediatric Rhinoconjunctivitis Quality of Life Questionnaire (PRQLQ) Score on Day 15 (Visit 4)
Description: The PRQLQ is a validated, disease-specific, quality-of-life (QOL) questionnaire developed to measure the physical, emotional, and social impairments that are experienced by children (aged ≥6 to <12 years) with rhinoconjunctivitis. The PRQLQ has 23 questions in 5 domains (nose symptoms, eye symptoms, practical problems, activity limitation and other symptoms). Subjects recall how they have been during the previous week and respond to each question on a 7-point scale with scores ranging from 6 (extremely bothered), 5 (very bothered), 4 (quite bothered), 3 (somewhat bothered), 2 (bothered a bit), 1 (hardly bothered at all), 0 (not bothered). The Overall PRQLQ score is the mean of all 23 subject-reported responses. The Overall PRQLQ score range from 0 to 6 where 0 represents no impairment and 6 represents maximum impairment.
Time Frame: Baseline and day 15
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GSP 301 NS | Placebo NS
Number analyzed (Participants) | 222 | 219
units on a scale
  Baseline | 2.51 (1.078) | 2.42 (1.001)
  Mean Change from baseline to end of treatment | -0.8 (0.08) | -0.5 (0.08)
Statistical Analysis 1: Comparison: GSP 301 NS vs Placebo NS; Test type: Superiority; p < 0.001, ANCOVA; Least Square Mean Difference = -0.3, 95% CI 2-sided [-0.5 to -0.1], Standard Error of Mean 0.09

4. Secondary Outcome: Change From Baseline in Average AM and PM Subject-reported 12-hour Reflective Total Ocular Symptom Score (rTOSS) Over the 14-day Treatment Period.
Description: The Total Ocular Symptom Score (TOSS) will be calculated using the 3 eye-related non-nasal symptoms: itching/burning eyes, tearing/watering eyes, and redness of eyes. The subject will assess and report his/her non-nasal symptoms twice (AM and PM assessments). Scores ranged from 0 (No sign/symptom evident), 1 (Sign/symptom clearly present but minimal awareness; easily tolerated), 2 (Definite awareness of sign/symptom that is bothersome but tolerable) and 3 (Sign/symptom is hard to tolerate; causes interference with activities of daily living and/or sleeping). The Total Ocular Symptom Score (TOSS) ranged from 0 to 9.
Time Frame: Baseline and day 14
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | GSP 301 NS | Placebo NS
Number analyzed (Participants) | 222 | 219
units on a scale
  Baseline | 3.84 (2.45) | 3.59 (2.52)
  Mean Change from baseline to end of treatment | -0.8 (0.14) | -0.6 (0.13)
Statistical Analysis 1: Comparison: GSP 301 NS vs Placebo NS; Test type: Superiority; p = 0.233, Mixed Models Analysis; Least Square Mean Difference = -0.2, 95% CI 2-sided [-0.6 to 0.1], Standard Error of Mean 0.19

ADVERSE EVENTS:
Time Frame: AEs and SAEs were collected from the time of signing the informed consent form (ICF) until the follow up contact which was approximately 22 days and up to 27 days with 7 to 10 days of a placebo run-in period and 14 days of treatment period, with allowable window periods for the study visits.
Arm/Group | GSP 301 NS | Placebo NS
All-Cause Mortality (participants affected / at risk) | 0/225 | 0/221
Serious Adverse Events (participants affected / at risk) | 0/225 | 1/221
Other Adverse Events (participants affected / at risk) | 0/225 | 0/221
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | GSP 301 NS (N=225) | Placebo NS (N=221)
Meningitis viral (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT03463031/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-06): https://cdn.clinicaltrials.gov/large-docs/31/NCT03463031/SAP_001.pdf